CLINICAL TRIAL: NCT05797597
Title: Long-term Aspirin Therapy as a Predictor of Decreased Susceptibility to SARS-CoV-2 Infection in Aspirin-Exacerbated Respiratory Disease
Acronym: AERD-CoV19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lucyna Mastalerz (Other)
Responsible Party: Sponsor-Investigator, Lucyna Mastalerz, Professor, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AERD-CoV19
Record Dates: First submitted 2023-03-01; First posted 2023-04-04 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: AERD - Aspirin Exacerbated Respiratory Disease
MeSH Terms: interventions — Aspirin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Experimental): Acard 300 mg (Acidum acetylsalicylicum). 1 tablet (300 mg) twice a day
  Interventions: Drug: Aspirin 300 Mg Oral Tablet
- Placebo (Placebo Comparator): Placebo 1 tablet twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin 300 Mg Oral Tablet — 8-week treatment of aspirin, then after 2-weeks washout the next treatment arm is placebo for 8 weeks
  Arms: Aspirin
Drug: Placebo — 8-week treatment of placebo, then after 2-weeks washout the next treatment arm is aspirin for 8 weeks
  Arms: Placebo

SUMMARY:
Aspirin-exacerbated respiratory disease (AERD) is characterized by the presence of asthma, chronic rhinosinusitis with nasal polyposis (CRwNP), and acute respiratory reactions induced by aspirin and other cyclooxygenase-1 inhibitors. One of the well-established therapeutic options is aspirin desensitization followed by daily aspirin therapy. The potential mechanisms underlying the clinical benefit of this approach include the downregulation of CysLT1 receptor, inhibition of PGD2 and interleukin IL-4 via the signal transducer and activator of transcription 6, global (blood, urine) activation of type 2 (T2) inflammation as well as local (sputum) reduction of T2 asthma inflammation. Indeed, among current aspirin-treated patients with AERD (n=37), no one had severe acute respiratory syndrome coronavirus clade 2 (SARS CoV-2) infection and most importantly, none of them developed COVID19 during pandemic. WHY? Notably, patients with AERD did not have asthma and nasal polyps exacerbation on aspirin, which is in line with other studies. Respiratory infections, such as the current COVID-19 pandemic, target epithelial cells in the respiratory tract. SARS-CoV-2 spike (S) protein binds angiotensin-converting enzyme 2 (ACE2), and in concert with host proteases, principally transmembrane serine protease 2 (TMPRSS2), promotes cellular entry. Nasal and bronchial epithelium play a key role in the early phases of an immune response to respiratory viruses. Induced sputum (IS) and nasal lavage (NL) cells are likely the first immune cells to encounter SARS CoV-2 during an infection, and their reaction to the virus will have a profound impact on the outcome of the infection. Interferons (IFNs) are antiviral cytokines and among the first mediators produced upon viral infection. IFNs are divided into three groups based on their receptor usage; type I IFNs (IFN-α and IFN-β), type II IFN (IFN-γ), and type III IFNs (IFN-λ1 and 2). Both production of IFN and cellular response to IFN are critical steps for the restriction of viral dissemination. An interferon-stimulated gene (ISG) is a gene whose expression is stimulated by interferon. Specifically, type I and type III interferons are antiviral cytokines, triggering ISGs that combat viral infections. The type II interferon class only has one cytokine (IFN-γ), which has some antiviral activity. To conclude, the assessment of gene expression for interferon α1 (IFNA1), interferon β1 (IFNB1), interferon γ (IFNG), interferon λ1 and λ2 (IFNL1 and IFNL2) as well as for ACE2 and TMPRSS2 in sputum and nasal cells may shed new light on the course of this infection in patient with AERD during long term aspirin therapy.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR AERD PATIENTS:

* signed informed consent form
* 18-70 years old AERD patients with baseline FEV1 of at least 70% of the predicted value on the challenge/desensitization day
* no pregnancy, higly effective contraception must be used

INCLUSION CRITERIA FOR HEALTHY CONTROL:

* signed informed consent form
* 18-70 years old and healthy condition
* no asthma

Exclusion Criteria:

* failure of the circulatory and respiratory system, liver, kidneys and other vital organs
* diabetes, cancer, systemic diseases of connective tissue, infectious diseases, coagulation disorders, active peptic ulcer disease, any active bleeding process.
* Use of drugs that interact with aspirin
* use of intoxicants, alcohol abuse, active and passive smoking,

  * pregnancy, lactation.
  * hypersensitivity to the active substance or any of the excipients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with two-fold decrease in gene expression of ACE2, TMPRSS2, BSG, PPIA, PPIB, DPP4, IFNA1, IFNB1 IFNG, IFNL1, IFNL2 and ISG in sputum and nasal cells after 8 weeks of placebo/aspirin therapy compared to the baseline value. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lucyna Mastalerz, prof., Principal Investigator — Jagiellonian University
Locations (1):
- University Hospital, Pulmunology Clinic, Krakow, Poland